CLINICAL TRIAL: NCT00911755
Title: Randomized Controlled Trial to Evaluate the Efficacy of Video-laryngoscopy vs. Direct Laryngoscopy for Endotracheal Intubation in the Critically Ill Patients: A Pilot Study
Brief Title: Videolaryngoscopy in the Critically Ill
Acronym: VICI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H08-02826
Record Dates: First submitted 2009-05-29; First posted 2009-06-02 (Estimated); Last update posted 2014-02-19 (Estimated); Status verified 2014-02

CONDITIONS: Endotracheal Intubation
Keywords: Laryngoscopy; Glidescope
MeSH Terms: interventions — Intubation, Intratracheal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Laryngoscopy (Other)
  Interventions: Procedure: Endotracheal Intubation
- Videolaryngoscopy (Other)
  Interventions: Procedure: Endotracheal Intubation

INTERVENTIONS:
Procedure: Endotracheal Intubation — This study is comparing 2 currently accepted methods of endotracheal intubation: laryngoscopy and videolaryngoscopy
  Arms: Laryngoscopy
Procedure: Endotracheal Intubation
  Arms: Videolaryngoscopy

SUMMARY:
Endotracheal Intubation (ETI) is done to place a plastic tube in a patient's trachea (windpipe) to assist with breathing. Patients admitted to the intensive care unit (ICU) are the sickest of patients and the majority of them require this life saving procedure. A critical illness can be sudden and ETI required urgently. The doctors performing ETI in these situations may not be experts at ETI. Studies have shown that if it takes more than one attempt to get the tube in the right position patients can have severe complications such as: decrease level of oxygen in the body, decrease blood pressure, and cardiac arrest. These complications can be life threatening and increase the length of time spent in an ICU.

To perform ETI the doctor uses a metal tool called a laryngoscope that is placed through the patient's mouth to open the throat and then pass the tube into the trachea. The type of procedure that has been used for many years is called Direct Laryngoscopy (DL) which means that the doctor looks through the mouth directly into the throat. Newer technology is available and can be used at VGH called Video Laryngoscopy (VL). With VL there is a camera on the end of the laryngoscope and a video image is displayed on a monitor making it easier to see the entrance to the trachea. VL is not available for all cases at VGH and is unavailable in many other hospitals.

In this study we will compare DL to VL. Patients will be randomly placed in one of two groups: first attempt at ETI done with DL or first attempt of ETI done with DL. Patients will only be considered eligible for this study if the doctor feels that either DL or VL would be appropriate for the patient. In this pilot study we hope show that conducting a larger study would be feasible. If a larger study were to show that VL decreases complications and shortens length of ICU stay we would be able to recommend this procedure for all ETI at VGH as well as other hospitals where it currently may not be available.

DETAILED DESCRIPTION:
Hypothesis: In this study, we hypothesize that videolaryngoscopy (VL) is associated with a decreased risk of intubation failure compared to direct laryngoscopy in the critically ill. We also hypothesize that VL is associated with fewer number of intubation attempts and decreased risk of complications compared to DL.

Background: In the critically ill, endotracheal intubation is a high-risk procedure with complications occurring in up to 54% of patients. Our own published work has demonstrated that more than one attempt at intubation occurred in 33% of patients and was associated with a three-fold increased risk of severe complications. VL provides a superior laryngeal view when compared to DL which may translate into less failed intubations, and resultant decreased complications.

Specific objectives:

1. Determine point estimates for failure to intubate on the first attempt, which can then be used to power a larger efficacy trial examining VL vs. DL in the critically ill.
2. Compare VL vs. DL on risk of intubation failure (as defined by one than more attempt)
3. Compare VL vs. DL on number of attempts at endotracheal intubation, time-to-intubate, and risk of complications.

Methods:

1. Design: Single center, randomized-controlled pilot study
2. Patients: Forty critically ill patients requiring urgent endotracheal intubation (within 30 minutes) by the intensive care team.
3. Intervention: Patients will be randomized to initial attempt at intubation by VL vs DL.
4. Power Calculation: Given this is a pilot study to generate point estimates, power calculations have not been performed. However, 20 patients in each arm will provide a robust point estimate that can be used to power a future efficacy study.
5. Analysis: Data will be analyzed in an intention-to-treat fashion. Our primary objective, failure to intubate on the first attempt, will be analyzed using Fisher's exact test. This test will also be used to analyze the risk of complications comparing VL to DL. Number of attempts at intubation and time-to-intubation will be analyzed using a Wilcoxon rank-sum test.
6. Potential Pitfalls: As slow recruitment is always a concern, we conservatively estimate that 5 patients will be enrolled per month, thus requiring a total of 8 months for patient accrual.

Significance: If VL results in fewer complications during endotracheal intubation, then this technique may become widely adopted for this high risk procedure. Furthermore, in many centers, anesthesiology support for airway management of the critically ill may be limited, if at all present. Thus, the impact of this research may be even more applicable outside of the tertiary teaching centers where airway management expertise is readily available.

ELIGIBILITY:
Inclusion Criteria:

* Any patient over the age of 16 years, requiring urgent (within 30 minutes) endotracheal intubation, who are attended to by the critical care team will be eligible for enrolment

Exclusion Criteria:

* Patients who require intubation within 5 minutes or have contraindications to either of the study intubation technique will be ineligible
* cardiac arrest
* cardiopulmonary instability (oxygen saturation <90% or systolic blood pressure < 80 mmHg despite oxygen or fluid therapy)
* any clinical deterioration while awaiting randomization
* known prior or anticipated difficult intubation
* need for awake intubation (defined by sedation, topicalization and avoidance of neuromuscular blockade)
* pregnancy
* cervical spine precautions
* any patient deemed inappropriate for enrolment by the attending physician

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2009-07; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
risk of failure on the first attempt of endotracheal intubation

SECONDARY OUTCOMES:
number of attempts at laryngoscopy
time to successful intubation
number of complications

CONTACTS AND LOCATIONS:
Overall Officials: Donald EG Griesdale, MD, Principal Investigator — University of British Columbia; P Choi, Study Director — University of British Columbia; G Isac, Study Director — University of British Columbia; V Dhingra, Study Director — University of British Columbia; A Chau, Study Director — University of British Columbia; C Menon, Study Director — University of British Columbia
Locations (1):
- Vancouver General Hospital, Intensive Care Unit, Vancouver, British Columbia, Canada

REFERENCES:
- [Derived] Griesdale DE, Chau A, Isac G, Ayas N, Foster D, Irwin C, Choi P; Canadian Critical Care Trials Group. Video-laryngoscopy versus direct laryngoscopy in critically ill patients: a pilot randomized trial. Can J Anaesth. 2012 Nov;59(11):1032-9. doi: 10.1007/s12630-012-9775-8. Epub 2012 Aug 30. PMID 22932944